CLINICAL TRIAL: NCT01567488
Title: A Phase II Study on Everolimus, an mTOR Inhibitor (Oral Formulation), With Octreotide LAR® in Adult Patients With Advanced, Non-functioning, Well-differentiated Gastrointestinal Neuroendocrine Tumours (GI NET)
Brief Title: Phase II Study of Everolimus Combined With Octreotide LAR to Treat Advanced GI NET
Acronym: EVERLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE 1003; CRAD001KES08T (Other Grant/Funding Number: Novartis Farmacéutica S.A.)
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-05

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Advanced; Non functioning; Well differentiated
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus + Octreotide LAR treatment (Experimental)
  Interventions: Drug: Everolimus; Drug: octreotide LAR

INTERVENTIONS:
Drug: Everolimus — Everolimus 10mg/day
  Other Names: Afinitor
Drug: octreotide LAR — 30 mg each 28 days
  Other Names: Sandostatin LAR

SUMMARY:
The underlying hypothesis of the synergistic activity of octreotide and everolimus is based on the combination of a) a direct action of everolimus over mTOR (mammalian target of rapamycin), and b) the inhibitory effect of octreotide on the IGF-I (insulin like growth factor 1) system preventing the activation of the mTOR system by this factor. Both types of inhibition would completely cancel this signal transduction pathway, which is so important in neuroendocrine tumours.

Furthermore, the biological study proposed in this protocol will allow for better establishing the relationship between the activation of the IGFR-PI3K-mTOR signal transduction pathway (i.e., the mTOR pathway stimulated by IGFR) and treatment response; this information is relevant since the IGFR-PI3K-mTOR activation status could be a response prediction factor.

This study will provide significant additional information about the efficacy of the combination treatment of everolimus with octreotide LAR® in non-functioning GI NET.

DETAILED DESCRIPTION:
Everolimus has been developed following two administration regimens: weekly and daily. Phase I pharmacodynamic studies recommend doses of 50 mg weekly and 10 mg/daily, based on its toxicity and inhibitory effect of the mTOR pathway in tumours; although the inhibition of this pathway has been demonstrated, the knowledge of response prediction factors has not been developed, in part due to the very low responses found in the population in phase I studies. These factors can be better outlined in a phase II study, where patients who have received fewer previous treatments can respond better, and where the profile of responders and non-responders can be identified more easily.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-operable or metastatic non-functioning, well differentiated advanced GI NET, confirmed by cytology or histology. In case of liver metastasis, neuroendocrine tumours of unknown origin are accepted.
* Confirmation of diagnosis of neuroendocrine carcinoma of low to intermediate histology grade
* Radiologically documented disease progression within 12 months prior to inclusion in the study. If the patient received anticancer treatment within the past 12 months, disease progression must be documented by radiology during or after taking this medication
* Adequate bone marrow. liver and renal function

Exclusion Criteria:

* Previous treatment with mTOR inhibitors (sirolimus, temsirolimus, everolimus, deforolimus).
* Patients with any serious disease and/or an uncontrolled clinical condition
* Patients on chronic treatment with corticosteroids or any other immunosuppressive agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06-08 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with progression-free survival (PFS) | After 12 month of study treatment
  Rate of patients

SECONDARY OUTCOMES:
Number of patients positive for insulin like growth factor 1 receptor (IGF1R) and ribosomal kinase S6 (S6K) phosphorylation. | At baseline
  Activation status of mTOR pathway.
Rate of patients with objective responses | Each three cycles
  Includes duration of response
Median and average of time for Overall survival | At the end of the study
  Time from inclusion date up to date of death for any reason.
Rate of patients with an early decrease of chromogranin A (CgA) levels | Each cycle
  CgA levels will be measured when increased at baseline and up to its normalization.
Percentage of patients with Adverse Events | Each cycle
  Ocurred during the trial and up to 30 days after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Salazar, MD, PhD, Study Chair — Grupo Espanol de Tumores Neuroendocrinos
Locations (1):
- Instituto Catalán de Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
As per Spanish local regulations

REFERENCES:
- [Derived] Capdevila J, Teule A, Barriuso J, Castellano D, Lopez C, Manzano JL, Alonso V, Garcia-Carbonero R, Dotor E, Matos I, Custodio A, Casanovas O, Salazar R; EVERLAR study investigators. Phase II Study of Everolimus and Octreotide LAR in Patients with Nonfunctioning Gastrointestinal Neuroendocrine Tumors: The GETNE1003_EVERLAR Study. Oncologist. 2019 Jan;24(1):38-46. doi: 10.1634/theoncologist.2017-0622. Epub 2018 May 23. PMID 29794066